CLINICAL TRIAL: NCT01250314
Title: Radiological, Biological, Genetic and Micro-architectural Bone Determinants of Fractures in Men With Low Bone Mineral Density
Brief Title: Radiological Biological Genetic and Micro-architectural Bone Determinants of Fractures in Men With Low Bone Mineral Density
Acronym: OSTEHOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: P070121
Record Dates: First submitted 2010-11-27; First posted 2010-11-30 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-07

CONDITIONS: Osteoporosis
Keywords: osteoporosis; men; bone micro-architecture; bone markers
MeSH Terms: conditions — Osteoporosis; Multiple Endocrine Neoplasia Type 1 | interventions — X-Rays; Biological Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With fracture (Other): Patients with fracture
  Interventions: Other: Radiology; Other: Biological, biochemical and genetic samples
- Without fracture (Other): Patients without fracture
  Interventions: Other: Radiology; Other: Biological, biochemical and genetic samples

INTERVENTIONS:
Other: Radiology — Spine radiography, densitometry, evaluation of bone architecture and micro-architecture (computed tomography of lumbar spine and hip and peripheral micro-scanner (XREME SCANCO) at tibia and wrist).
Other: Biological, biochemical and genetic samples — *Serum calcium and phosphore evaluation, bone remodeling markers, 25-hydroxyvitamin D level assessment: Blood samples plasma (5 ml):Creatin, calcemia, phosphoremia, alkaline phosphatase, bone alkaline phosphatase, osteocalcin, CTX, 25 hydroxyvitamin D and parathormone
  Urinary samples :
  Deoxy-pyridinoline, creatinuria Fasting morning urine on a sample Calciuria, creatinuria, cortisoluria Day urine on a sample
  *Assessment of possible determinants of fractures in man
  Blood samples plasma (5 ml):
  * Sexual Hormones: Estradiol, Testosterone, SHBG, LH, FSH
  * Homocysteine
  * IGF1
    * Extraction of DNA for a genetic polymorphism study:
  Sample of 10 ml of blood on EDTA for DNA extraction.
  Tested polymorphisms will be: LRP5, CYP19 (Aromatase), COL1A1 (Collagen I),MHTFR, IGF-1,VDR vitamin D receptor
  Globally 20 ml of blood will be taken for each subject. Every biological sample for biochemical dosages and for genetic analysis will be preserved in an anonymous way.

SUMMARY:
Rational: Osteoporosis in men is responsible for one third of fragility fractures. However the definition and especially the determinants of fracture in humans are less well known than in women.

Primary Objective: To search radiologic, biochemical, genetic and micro-architecture bone factors associated to fractures in men with low bone density.

Study design: case/control study (fracture vs. no fracture) with men selected according to low bone density (Z-score<-2).

Eligibility criteria: Included subjects will be men whose age is ³ 40 and £ 70 years with a Z-score< -2 at least at one of the 3 measured sites (wrist, lumbar spine, femoral neck). Subjects with secondary osteoporosis will be excluded (corticosteroid treatment, hypogonadism, …) Progress of the study: The recruitment will be over two years. The study will include two periods, an inclusion visit and a period of 3 months to achieve radiological and biological examinations. The subjects will be recruited in the 3 rheumatology departments (LARIBOISIERE, COCHIN). Subjects will be investigated at LARIBOISIERE hospital to perform radiological examinations and biological sampling for laboratory tests within 3 months of enrollment.

Evaluation criteria: Biochemistry: dosages of sexual steroids, bone remodeling markers and homocysteine; Genetic: evaluation of polymorphism of candidates genes associated to fragility fractures (collagen type I, homocysteine, LRP5); Radiology: evaluation of bone micro-architecture with a scan of lumbar spine and hip and peripheral micro-scan (XTREME sSCANCO) and bone densitometry at spine, femoral neck and wrist.

Duration of participation: there is no follow up Total duration of the study: 2 years and 3 months. Number of subjects: 100 patients with fracture and 100 controls without fracture

DETAILED DESCRIPTION:
Statistical Analysis: Relationship between computed scan parameters at different sites, bone micro-architectural parameters (peripheral scan), biological parameters, genetic markers and the occurrence of fracture will be analyzed initially by univariate analysis (screening process). This will help to reduce the number of variables analyzed at the second stage of analysis (i.e. multivariate analysis).

Expected results: This study will help to evaluate radiological, biochemical and genetic determinants of bone quality in men with decreased bone density. It will help to establish a prospective study to evaluate predictive factors of fractures in men.

ELIGIBILITY:
Inclusion Criteria:

* Subject of masculine gender
* Aged ≥ 40 years and ≤ 70 years
* Subject with Z-score < -2 at least one of 3 sites
* one of 3 sites (wrists, lumbar spine (defined on at least 2 continuous evaluable vertebrae between L1-L4) and femoral neck) discovered incidentally or not
* Subject who have signed the informed consent form

The inclusion densitometry examination, less than 6 months old, will be performed on a Lunar or Hologic system. The reference data are the French reference data included in the Lunar system and TK in the Hologic system).

Exclusion criteria:

* Patient or control subject with no affiliation at health national system (beneficiary or co-beneficiary)
* Subject who received any corticoid treatment more than 3 months along
* Subject with any known seropositivity for HIV
* Subject with a chronic inflammation disease (rheumatoid polyarthritis, ankylosing spondylarthritis, inflammatory bowel)
* Subject with secondary osteoporosis documented by clinical and biological examinations (serum calcium, serum phosphate, serum phosphatase alkaline, gamma GT, testosterone) in order to eliminate any chronic alcoholism, alcoholic cirrhosis, hypogonadism, osteomalacia, hemochromatosis, hyperthyroidism, primitive hyperparathyroidism, hypercorticism
* Subject who received treatment with bisphosphonates intravenously
* Subject who received a treatment with bisphosphonates (Actonel® or Fosamax®) for at least 5 years and stopped since less than 2 years
* Subject who received a treatment with bisphosphonates for at least 3 years and stopped since less than 1 year
* Subject who received a treatment with bisphosphonates during the 6 months before inclusion

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2008-02; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Biochemical | up to 90 days
  Sexual steroid dosages, bone remodeling markers, homocysteine, IGF1
Genetic | up to 90 days
  Polymorphism evaluation of candidate genes associated to fractures of fragility (collagen type I, receptor of 25-hydroxy vitamin D, aromatase, MTHFR, LRP5)
Radiological | up to 90 days
  Bone micro-architecture evaluation with a scanner examination of lumbar spine and hip, peripheral scanner (Xtreme Scanco) and bone mineral densitometry at spine, femoral neck and wrist.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Christine De VERNEJOUL, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Fédération de Rhumatologie - Hôpital LARIBOISIERE, Paris, France